CLINICAL TRIAL: NCT02534324
Title: The Effect of Pre-discharge Blood Pressure on the Follow-up Outcomes After Managing the Patients With Asymptomatic Severe Hypertension in Emergency Department
Brief Title: The Effect of Pre-discharge Blood Pressure of Patients With Asymptomatic Severe Hypertension in Emergency Department
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khrongwong Musikatavorn, MD., Dr., Chulalongkorn University
Other Study IDs: 397/57
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension; Emergencies; Asymptomatic Conditions
Keywords: Hypertension; Emergency
MeSH Terms: conditions — Hypertension; Emergencies; Asymptomatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High SBP+antihypertensive meds: Patients with pre-discharge systolic blood pressure at discharge < 180 mmHg
  Interventions: Drug: Antihypertensive meds
- Severely high SBP+antihypertensive meds: Patients with pre-discharge systolic blood pressure at discharge >= 180 mmHg
  Interventions: Drug: Antihypertensive meds

INTERVENTIONS:
Drug: Antihypertensive meds — Antihypertensive medications will be given to newly-diagnosed or non-compliant cases. The additional oral antihypertensive drugs instruction to adjust their current regimens will be given to the patients with underlying hypertension for more BP control. The choices of drugs will be at discretion of treating physicians.
  Other Names: Blood pressure-lowering drugs

SUMMARY:
The current guideline of asymptomatic severe hypertension (ASH) treatment in emergency department (ED) recommends through low level of evidence that the patients should not be rapidly decreased their BP in ED but instead receive oral antihypertensive treatment and close outpatient follow-up is needed. Unfortunately, there was some ambiguity in the time point of BP measurement in ED described in the past literature because high BP on ED admission may significantly decrease within hours without any medications. The importance of pre-ED discharge BP, which can still be critically high, that may affect the follow-up outcome has never been investigated. The study aim of this study is to evaluate the physicians' treatment strategies as well as immediate clinical outcomes between patients with severely- and moderately-elevated pre-discharge BP after management of ASH its in ED during the recent recommendation. The secondary outcome is to compare the BP at follow-up in these two groups.

DETAILED DESCRIPTION:
The investigators will follow the patients with asymptomatic severe hypertension who attend ED of King Chulalongkorn Memorial Hospital (KCMH), an urban, 1,500-bed, university-affiliated, tertiary care hospital as well as treatment strategies. A management strategy whether to start the drugs in ED with or without a period of observation or immediately after discharge without any observation depends on the treating physicians' judgment. The investigators predefined the pre-discharge BP at ED into two groups; high BP (pre-discharge SBP < 180 mmHg) and severely high BP (pre-discharge SBP >= 180mmHg) groups. Every eligible patient was scheduled for the internal medicine clinic for continuous care of the high blood pressure within 3-7 days after discharge. Medical records were retrieved for the follow-up BP, compliance and associated adverse events at the clinic. The investigators will make telephone follow-ups to the participants or their contact personnel in every case at 10 days after ED presentation to identify the deceased cases or those with major morbidity as well as the compliance to their medications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old
* Systolic BP (SBP) greater or equal to 180 mmHg
* Diastolic BP (DBP) ≥ 100 mmHg

Exclusion Criteria:

* Acute end-organ damage related to severe hypertension that required rapid intravenous antihypertensive drugs for acute treatment involving cardiovascular (acute chest pain, heart failure, acute coronary syndromes, acute aortic syndromes), renal (acute kidney injury), ocular (retinal hemorrhage or hypertensive retinopathy) and central nervous system (seizure, acute cerebrovascular diseases, hypertensive encephalopathy)
* Hypertension caused by medical toxicology (e.g. use of sympathomimetic drugs (amphetamine and its derivatives), alcohol withdrawal syndrome
* Significantly decreased renal function (serum creatinine ≥ 1.5 mg/dL or creatinine clearance ≤ 30 ml/min)
* Pregnant women
* Moderate to severe pain (pain score on visual analog scale ≥ 5 centimeters out of 10)
* BP decrease to less than 180 mmHg after 10-minute bed rest without any medical treatment
* Having concurrent medical conditions that needed hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) who presented in our ED with systolic BP (SBP) greater or equal to 180 mmHg and diastolic BP (DBP) ≥ 100 mmHg were consecutively enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khrongwong Musikatavorn, M.D., Principal Investigator — Faculty of Medicine, Chulalongkorn Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Patumwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakprasert P, Musikatavorn K, Rojanasarntikul D, Narajeenron K, Puttaphaisan P, Lumlertgul S. Effect of predischarge blood pressure on follow-up outcomes in patients with severe hypertension in the ED. Am J Emerg Med. 2016 May;34(5):834-9. doi: 10.1016/j.ajem.2016.01.013. Epub 2016 Jan 21. PMID 26874395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients >= 18 years old who presented in ED with systolic BP >=180 mmHg and diastolic BP >= 100 mmHg were enrolled. The patients with minor chief complaints that were not related to severe hypertension or those who presented to hospital for routine outpatient visits and were referred to ED due to severe hypertension were included.
Period: Overall Study
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds
Started | 98 | 48
Completed | 73 | 40
Not Completed | 25 | 8
Not completed — Protocol Violation | 4 | 1
Not completed — Lost to Follow-up | 20 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds | Total
Number analyzed (Participants) | 98 | 48 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (15.1) | 64.2 (15.0) | 64.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 27 | 89
  Male | 36 | 21 | 57
Region of Enrollment [Number; unit: participants]
  Thailand | 98 | 48 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died Within 7 Days After Discharge From the Emergency Department
Description: Number of participants who died from hypertension-related events within 7 days after discharge from the emergency department.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds
Number analyzed (Participants) | 98 | 48
participants | 0 | 0

2. Secondary Outcome: Number of Participants Who Had Major Hypertensive-related Events After Discharge From the Emergency Department
Description: Participants who had major hypertensive-related events defined by those who had one or more of the followings: acute chest pain, heart failure, acute coronary syndromes, acute aortic syndromes, retinal/vitreous hemorrhage, hypertensive retinopathy, seizure, acute cerebrovascular diseases, hypertensive encephalopathy, which occurred within 7 days after discharge from emergency department.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds
Number analyzed (Participants) | 98 | 48
participants | 1 | 0
Statistical Analysis 1: Comparison: High SBP+Antihypertensive Meds vs Severely High SBP+Antihypertensive Meds; Test type: Superiority or Other; p = 0.49, Chi-squared

3. Secondary Outcome: Systolic Blood Pressure at Follow-up
Description: Systolic blood pressure at follow-up measured by physicians that were non-investigators and unaware of the study.
Time Frame: 3 to 7 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds
Number analyzed (Participants) | 73 | 40
mmHg | 153.7 (25.7) | 160.9 (23.0)
Statistical Analysis 1: Comparison: High SBP+Antihypertensive Meds vs Severely High SBP+Antihypertensive Meds; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | High SBP+Antihypertensive Meds | Severely High SBP+Antihypertensive Meds
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/48
Other Adverse Events (participants affected / at risk) | 0/98 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High SBP+Antihypertensive Meds (N=98) | Severely High SBP+Antihypertensive Meds (N=48)
Aortic aneurysm (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The results may not be generalizable to other centers with different treatment practices. We still had a considerable percentage of patients who were lost-to-follow-up that may have affected the results. The size of population was relatively small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes